CLINICAL TRIAL: NCT02049892
Title: A Comparison of Large Diameter Metal Heads vs. Small Diameter Metal Heads vs/ Dual Mobility Total Hip Replacements
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert T. Trousdale, PI, Mayo Clinic
Other Study IDs: 13-002050
Record Dates: First submitted 2014-01-22; First posted 2014-01-30 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Total Hip Replacement
Keywords: Total Hip Replacement; Metal Ion; 2-5 years after surgery; Asymptomatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metal Ion
  Interventions: Other: Metal Ion Levels

INTERVENTIONS:
Other: Metal Ion Levels

SUMMARY:
Does having a large diameter metal on polyethylene total hip replacement increase metal ion release. Larger metal heads are thought to have increased torsional forces on the trunion which would like release more metal ions. Increased metal ion levels have been associated with adverse local tissue reactions. Are there any differences comparing these groups to a dual mobility type total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* One total hip replacement, either a large metal head (>40) or a small metal head (<30) on a polyethylene bearing surface.
* 2 to 5 years s/p surgery minimum. No symptoms

Exclusion Criteria:

* Any other bearing surface besides metal on poly, no other joint replacements, symptomatic

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic patients with prior hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-12-01; Primary Completion 2016-01-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Metal Ion levels | 2 years
  We would like to determine a difference in metal ion levels on metal on polyethylene total hip replacement

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States